CLINICAL TRIAL: NCT06078319
Title: Ruxolitinib Adherence in Myelofibrosis and Polycythemia Vera
Acronym: RAMP
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: 1064/2020/Oss/AOUBo
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-02

CONDITIONS: Adherence, Patient; Adherence, Treatment
MeSH Terms: conditions — Patient Compliance; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prospective multicenter observational cohort study will be offered consecutively to any patient with primary or secondary myelofibrosis or with Polycythemia Vera who has initiated therapy with ruxolitinib, prescribed as part of the normal course of care and completely independent of study participation. The main purpose is to assess adherence to ruxolitinib using the ARMS questionnaire. Each individual patient will be administered the questionnaire at the first convenient opportunity, regardless of when ruxolitinib is started, and again after 4, 8, 12, 24, and 48 weeks, in conjunction with drug procurement.

DETAILED DESCRIPTION:
The prospective multicenter observational cohort study will be offered consecutively to any patient with primary or secondary myelofibrosis or with Polycythemia Vera who has initiated therapy with ruxolitinib, prescribed as part of the normal course of care and completely independent of study participation. Laboratory tests and histologic, cytogenetic, molecular, and radiologic investigations performed by the patient and collected for study will be conducted in accordance with clinical practice, independent of the patient's participation in the study. In particular, data related to systemic symptoms and splenomegaly will be collected at diagnosis and disease reassessments performed in the context of normal clinical practice. These data will be collected at the first administration of the ARMS questionnaire and again after 12, 24, and 48 weeks. If performed, any additional assessments will also be recorded. Each individual patient will be administered the questionnaire (ARMS) at the first convenient opportunity, regardless of the time of initiation of ruxolitinib, and again after 4, 8, 12, 24, and 48 weeks, in conjunction with drug procurement. If in-person data collection is not possible, the mode of data collection by telephone interview will be adopted. The minimum expected duration of individual patient observation is 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients diagnosed with Primary Myelofibrosis or secondary to Essential Thrombocythemia/Polycythemia Vera or diagnosed with Polycythemia Vera who are in the treatment with ruxolitinib therapy in accordance with normal clinical practice
* Obtaining informed consent for data collection and processing
* The Patient must come to the in-person visit at least once, an occasion on which informed consent to 'study membership will be offered

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary MF or secondary to Essential Thrombocythemia/PV or diagnosed with PV, aged 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence | 2 years
  Incidence of low adherence to ruxolitinib therapy, and the features associated with low adherence
Distress | 2 years
  Emotional distress is measured based on a visual analogue scale with the distress thermometer, a simple and quick (3-4 minutes) tool that investigates the areas most involved in distress (minimum value: 0, lower distress; maximum value: 10, higher distress)

CONTACTS AND LOCATIONS:
Locations (28):
- Italy (28):
  - Azienda Ospedaliera Annunziata, Cosenza, Calabria
  - Grande Ospedale Metropolitano "Bianchi Melacrino Morelli", Reggio Calabria, Calabria
  - Università degli Studi di Napoli Federico II - U.O.C. di Ematologia e Trapianti di midollo, Napoli, Campania
  - IRCCS Policlinico Sant'Orsola, Bologna, Emilia-Romagna
  - Università degli studi di Ferrara - Nuovo Polo Ospedaliero di Cona - A.O.U. Arcispedale S. Anna, Ferrara, Emilia-Romagna
  - Azienda Ospedaliero-Universitaria di Parma, Parma, Emilia-Romagna
  - AUSL di Piacenza - Palazzine Medicine Specialistiche, Piacenza, Emilia-Romagna
  - Dipartimento Oncoematologico - AUSL della Romagna, Ravenna, Emilia-Romagna
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - A.O.U. Integrata di Udine, Udine, Friuli Venezia Giulia
  - Ospedale S. Eugenio, Rome, Lazio
  - A.O.U. Policlinico Umberto I - Università degli Studi di Roma "La Sapienza", Rome, Lazio
  - Ospedale Belcolle, Viterbo, Lazio
  - IRCCS Azienda Ospedaliera Universitaria "San Martino" - IST, Genoa, Liguria
  - ASST Spedali Civili di Brescia, Brescia, Lombardy
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Gerardo, Monza, Lombardy
  - Ospedale San Luigi Gonzaga, Orbassano, Piedmont
  - Department of Oncology, University of Torino, Turin, Piedmont
  - A.O.U. Città della Salute e della Scienza - Presidio Molinette, Turin, Piedmont
  - A. O. Ordine Mauriziano di Torino, Turin, Piedmont
  - Ospedale "A. Businco" - Dipartimento Scienze Mediche e Sanità Pubblica Università degli Studi di Cagliari, Cagliari, Sardinia
  - A.O.U. "Policlinico-V. Emanuele"- P.O. Ferrarotto, Catania, Sicily
  - A.O. Ospedali Riuniti Marche Nord - Presidio Ospedaliero San Salvatore, Pesaro, The Marches
  - Policlinico S.Maria alle Scotte, Siena, Tuscany
  - AOU di Padova, Padua, Veneto
  - A.O.U. Integrata Verona - Borgo Roma, Verona, Veneto